CLINICAL TRIAL: NCT00005883
Title: A Phase I - Part B Multiple Dose Trial of Phenethyl Isothiocyanate
Brief Title: Phenethyl Isothiocyanate in Preventing Lung Cancer in People Who Smoke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: CDR0000067923; P30CA016087 (NIH); NYU-9905; NCI-P00-0151
Record Dates: First submitted 2000-06-02; First posted 2004-04-28 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — phenethyl isothiocyanate

INTERVENTIONS:
Drug: phenethyl isothiocyanate

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. Phenethyl isothiocyanate may be effective in preventing lung cancer in smokers.

PURPOSE: Phase I trial of phenethyl isothiocyanate in preventing lung cancer in people who smoke.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of oral phenethyl isothiocyanate in smokers. II. Measure the steady state pharmacokinetics of phenethyl isothiocyanate required to maintain a steady state of this substance during the hours of 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK) exposure in these patients. III. Obtain preliminary data on the perturbation of NNK metabolism by phenethyl isothiocyanate in these patients.

OUTLINE: Patients complete a questionnaire containing a smoking and dietary log to assess cigarette and cruciferous vegetable consumption. Patients receive phenethyl isothiocyanate orally 4 times a day for 30 days. Cohorts of 3-6 patients receive escalating doses of phenethyl isothiocyanate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities. Patients are followed on days 35, 36, and 43.

PROJECTED ACCRUAL: A total of 15-27 patients will be accrued for this study over 4-6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Asymptomatic smokers who either refuse to or cannot stop smoking Urinary cotinine levels greater than 100 ng/mL Willing to adhere to certain dietary restrictions limiting intake of cruciferous vegetables (watercress, broccoli, radishes, mustard, brussels sprouts) while on study

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.6 mg/dL Transaminases less than 2 times normal Renal: Creatinine less than 1.6 mg/dL Urinary RBC levels 0-2 Urinary WBC levels at least 0-2 Pulmonary: No dyspnea at rest Other: No concurrent illness, condition, or symptom that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Primary Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Liebes, PhD, Study Chair — NYU Langone Health